CLINICAL TRIAL: NCT04099069
Title: The Impacts of the Different Anesthesia Methods on Patients of Transbronchial Cryobiopsy:A Prospective, Randomized, Controlled Trial
Brief Title: The Impacts of the Different Anesthesia Methods on Patients of Transbronchial Cryobiopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Director of the Respiratory department, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TS20180110
Record Dates: First submitted 2019-05-28; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Transbronchial Cryobiopsy; Anesthesia; Tracheal Intubation; Rigid Bronchoscopy; Safety
Keywords: Transbronchial Cryobiopsy; anesthesia; tracheal intubation; rigid bronchoscopy; safety; interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trachial intubation (Placebo Comparator): patient was insert trachial intubation with normal frequency jet ventilation
  Interventions: Procedure: anesthesia
- rigid bronchoscopy (Experimental): patient was insert trachial intubation with high frequency jet ventilation
  Interventions: Procedure: anesthesia

INTERVENTIONS:
Procedure: anesthesia — patient was insert trachial intubation or rigid bronchoscopy with ventilation under general anesthesia
  Other Names: insert rigid bronchoscopy under general anesthesia

SUMMARY:
to evaluate the difference between the tracheal intubation (TI) and rigid bronchoscopy (RB) under general anesthesia on patients with transbronchial cryobiopsy.

DETAILED DESCRIPTION:
To evaluate the difference between the tracheal intubation (TI) and rigid bronchoscopy (RB) under general anesthesia on patients with transbronchial cryobiopsy. Comparing the difference between two groups in the operating duration, extubation duration, total anesthesia time, heart rate, blood pressure and arterial blood gas analysis. This is a prospective, randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are admitted in the institution as ILD, while undefined after thorough history collection, laboratory examination and radiological data.
2. Transbronchial cryobiopsy(TBCB) is indicated by clinicians for definitive diagnosis and patients are content with the examination with agreement signed.
3. Blood gas analysis, routine blood test, ECG examination, coagulation function, immunological examination, chest HRCT, and liver/kidney function test have been completed

Exclusion Criteria:

1. The radiological data indicates non-ILD
2. The clinical examinations mentioned above are not completed.
3. The patient cannot endure or does not agree the procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
the fluctuation of heart rate | 24 hours
  fluctuation of heart rate during the procedure
the fluctuation of blood pressure | 24 hours
  the fluctuation of blood pressure during the procedure
the fluctuation of arterial partial pressure of carbon dioxide | 24 hours
  the fluctuation of arterial partial pressure of carbon dioxide during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The first affilliated hospital of Guanghzhou Medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No